CLINICAL TRIAL: NCT06631976
Title: Comparison of Conservative Treatment Methods for Sleep Disorders, Pain, and Shoulder Function in Patients With Supraspinatus Tendon Injury.
Brief Title: Conservative Treatment in Patients With Supraspinatus Tendon Injury.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Lodz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RCT-Physio-Injections-4-groups
Record Dates: First submitted 2024-10-03; First posted 2024-10-08 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-10

CONDITIONS: Supraspinatus Injury; Sleep Disturbance
MeSH Terms: conditions — Parasomnias | interventions — Methylprednisolone Acetate; Rehabilitation; Nerve Block; Lidocaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Rehabilitation (Active Comparator): Rehabilitation Treatment - a group of patients will be treated using a standardized rehabilitation protocol.
  Interventions: Other: Rehabilitation
- Steroid (Experimental): Rehabilitation treatment combined with a subacromial corticosteroid injection. Patients will receive 1ml of methylprednisolone acetate (40mg/ml) into the subacromial-subdeltoid bursa.
  Interventions: Drug: 1ml of Depo-Medrol® injection; Other: Rehabilitation
- PRP (Experimental): Rehabilitation treatment combined with PRP injection. Patients will have an 11ml venous blood sample taken. After centrifugation, the obtained preparation will be administered to the patients intratendinously.
  Interventions: Other: Rehabilitation; Drug: Tropocells® PRP injection
- Nerve Block (Experimental): Rehabilitation treatment combined with suprascapular nerve block. Patients will receive 4ml of 2% lidocaine around the suprascapular nerve.
  Interventions: Other: Rehabilitation; Drug: Nerve block with 4ml of 2% lidocaine

INTERVENTIONS:
Drug: 1ml of Depo-Medrol® injection — 1ml of methylprednisolone acetate (40mg/ml) injection into subacromial bursa.
  Arms: Steroid
Other: Rehabilitation — Rehabilitation
Drug: Nerve block with 4ml of 2% lidocaine — Nerve block with 4ml of 2% lidocaine around the suprascapular nerve
  Arms: Nerve Block
Drug: Tropocells® PRP injection — Tropocells® PRP injection. Patients will have an 11ml venous blood sample taken. After centrifugation, the obtained preparation will be administered to the patients intratendinously.
  Arms: PRP

SUMMARY:
Rotator cuff injuries are a major cause of severe pain, often significantly impacting patients' sleep quality. For patients waiting for surgery or those not eligible for operative treatment, conservative treatment is recommended. In cases of minor injuries, physiotherapy is as effective as surgical intervention.

The aim of this study is: (1) to compare the speed, effectiveness, and durability of four implemented interventions in improving sleep quality, pain, and shoulder function, (2) to select the most optimal form of conservative treatment for patients with shoulder pain affecting sleep quality, and (3) to evaluate the expression of brain-derived neurotrophic factor (BDNF) and proBDNF (precursor) at the mRNA protein level before the planned intervention (T0), 1 month (T1), 3 months (T3), and 6 months (T6) after intervention.

The study results can assist physicians and physiotherapists in providing patients with therapy that not only relieves pain and improves function but also augments sleep quality, an aspect often overlooked in the literature yet greatly impacting patients' quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic partial incomplete thickness tear of the supraspinatus tendon, with a length below 1 cm and not exceeding 50% of the tendon thickness, confirmed by ultrasound examination.
2. Sleep disturbance symptoms for at least 1 month due to shoulder pain - PSQI score > 5.
3. Shoulder pain disrupting the quality of sleep.
4. BMI < 30.
5. Age 40-75.

Exclusion Criteria:

1. Other accompanying pain symptoms.
2. History of shoulder surgery.
3. Coexistence of psychiatric or neurological disorders.
4. Presence of comorbidities that may disrupt sleep.
5. Presence of risk factors impairing tissue regeneration and increasing the likelihood of injury progression - osteoporosis, diabetes, hypercholesterolemia.
6. Alcohol dependence, nicotine addiction, passive smoking.
7. Taking antibiotics from the fluoroquinolone group, sleep-affecting medications (such as melatonin, trazodone, zolpidem), antidepressants, antipsychotics, anxiolytics.
8. Lack of patient consent, lack of cooperation, or impaired verbal-logical communication.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-06-04 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Constant-Murley Score | 6 months
  The CMS is a widely used clinical assessment tool in orthopedics, specifically for evaluating shoulder function and outcomes following shoulder surgery or injury. The CMS comprises a set of objective and subjective measures to assess various aspects of shoulder function, including pain, range of motion, strength, and activities of daily living. These components are evaluated through a combination of patient-reported outcomes and physical examination by a healthcare professional.
Numeric pain Rating Scale | 6 months
  The NRS is a commonly used tool in clinical studies to assess pain intensity. It involves asking the patient to rate their pain on a scale from 0 to 10, with 0 indicating no pain and 10 indicating the worst possible pain.
Range of motion measurements | 6 months
  The assessment of the range of motion of the upper limb (shoulder) is a standard procedure used to evaluate the function and mobility of the shoulder joint. This assessment involves examining the range of motion in various directions, including flexion, extension, abduction, adduction, external rotation, and internal rotation.
Strength measurements | 6 months
  The assessment of upper limb muscle strength using a dynamometer is a standard procedure used to measure the force exerted by the muscles of the shoulder and arm. This assessment involves using a handheld dynamometer to quantify the maximum force produced during specific muscle actions. Muscle strength measurement will be conducted during movements of flexion, extension, and external and internal rotation with the arm adducted and abducted.
BDNF and proBDNF Assessment | 6 months
  BDNF belongs to a family of proteins called neurotrophins, which act through tyrosine kinase receptors, influencing nerve cells. They exert a neuroprotective effect by stimulating neurogenesis and neuroplasticity processes. In the context of sleep disorders, BDNF may influence the structural stability of neurons in brain areas related to sleep regulation, such as the hippocampus or prefrontal cortex. Disruptions in the balance of this protein may contribute to various sleep disorders. Increased expression of this protein may also contribute to disturbances in normal neuronal processes.
Pittsburgh Sleep Quality Index | 6 months
  The PSQI is a self-assessment questionnaire that evaluates seven different aspects of sleep in adults. It assesses parameters of sleep quality such as difficulty with falling asleep, problems with maintaining sleep continuity, daytime functioning, and questions regarding the most common causes of sleep disturbances in the past four weeks. All of these contribute to a score rated from 0 to 21 points. Scores higher than 5 points indicate low sleep quality and differentiate patients into 'poor' and 'good' sleepers. A validated Polish version of the PSQI will be utilized in the study.

SECONDARY OUTCOMES:
The Laitinen Pain Scale | 6 months
  The Laitinen Pain Scale, also known as the Laitinen Analogue Scale, is a pain assessment tool used in clinical settings to measure pain intensity. The questionnaire provides a quantitative measure of pain intensity, allowing healthcare providers to track changes in pain over time and assess the effectiveness of pain management interventions. It also facilitates communication between patients and clinicians, enabling more accurate pain assessment and tailored treatment plans.
The Simple Shoulder Test | 6 months
  The SST is a clinical assessment tool used to evaluate shoulder function and disability. The SST consists of 12 questions that assess the patient's ability to perform various shoulder-related activities of daily living. These activities include reaching overhead, reaching behind the back, and lifting objects. Each question is scored on a dichotomous scale (yes/no), with a score of 1 assigned for each activity the patient can perform without difficulty.
The American Shoulder and Elbow Surgeons | 6 months
  The ASES is a widely used clinical assessment tool designed to evaluate shoulder function and assess outcomes following treatment for various shoulder conditions. The ASES Shoulder Score comprises two main components: pain and function. The function component evaluates the patient's ability to perform various shoulder-related activities of daily living.
Supraspinatous muscle echogenicity measurement | 6 months
  The echogenicity of supraspinatus muscle and trapezius muscle will be determined using ImageJ software (National Institutes of Health, U.S.; https://imagej.nih.gov/ij/). The echogenicity ratio of supraspinatus/trapezius muscle will be calculated.
The assessment of the degree of fatty infiltration of the supraspinatus muscle | 6 months
  A 3-point scale with the echogenicity of the trapezius muscle serving as reference: grade 1, isoechogenic; grade 2, mildly hyperechogenic; grade 3, markedly hyperechogenic.
The Montreal Cognitive Assessment | 6 months
  The MoCA is a widely used screening tool designed to assess various cognitive domains, including attention, memory, language, visuospatial abilities, executive function, and orientation. The MoCA consists of a series of tasks and questions that evaluate different aspects of cognitive function. These include tasks such as naming a series of animals, remembering a list of words, drawing a clock face, and performing serial subtraction.
The Trail Making Test | 6 months
  The Trail Making Test is a neuropsychological test of visual attention and task switching. It has two parts, in which the subject is instructed to connect a set of 25 dots as quickly as possible while maintaining accuracy.[1] The test can provide information about visual search speed, scanning, speed of processing, mental flexibility, and executive functioning.
A 3D measurement of the Supraspinatus Injury | 6 months
  Measurement of the size of the injury in three planes: depth, width and length.
Ellman Classification of Partial-Thickness Rotator Cuff Tears | 6 months
  A scale which classifies an injury depending on the localization and size: Grade 1: Partial tear <3mm in depth, Grade 2: Partial tear 3-6 mm in depth, depth does not exceed half the thickness of the tendon from the tubercle to the joint. Grade 3: Partial tear >6mm in depth, depth exceeds half the thickness of the tendon from the tubercle to the joint. Full recovery will be defined as Grade 0. A: Articular sided; B: Bursal sided; C: Intratendinous
Athens Insomnia Scale | 6 months
  The questionnaire consists of 8 questions designed to assess insomnia. The first five questions align with the ICD-10 criteria for diagnosing insomnia, including assessments of difficulties with sleep onset, awakening, total sleep time, and overall sleep quality. The last three questions assess the daytime consequences of insomnia, such as mood, functioning, and daytime sleepiness. Each question is rated from 0 to 3 points, corresponding to 'no problem' or 'very serious problem,' respectively. In total, all assessed items yield a score of 24 points. A validated Polish version of the AIS will be used in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Michał Kanak, MD, Study Chair — Medical University of Lodz; Marcin Domżalski, Prof., Study Chair — Medical University of Lodz
Locations (1):
- Medical University of Lodz, Lodz, Łódź Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided
Undecided.